CLINICAL TRIAL: NCT02483871
Title: Dose Optimization of Rosuvastatin in Early Stage and Metastatic Estrogen Receptor Positive Breast Cancer Patients on Endocrine Therapy
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Enrollment did not meet anticipated goals. Eligibility was a challenge.
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00062343
Record Dates: First submitted 2015-06-25; First posted 2015-06-29 (Estimated); Last update posted 2017-06-05 (Actual); Status verified 2017-06

CONDITIONS: Breast Cancer
Keywords: Estrogen Receptor Positive
MeSH Terms: conditions — Breast Neoplasms | interventions — Rosuvastatin Calcium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Rosuvastatin (Experimental): Two Cohorts, one at 20 mg and one at 40 mg will enroll in a dose escalation of rosuvastatin
  Interventions: Drug: Rosuvastatin

INTERVENTIONS:
Drug: Rosuvastatin
  Other Names: Crestor

SUMMARY:
Patients will be treated in a dose escalation scheme to investigate a role for the addition of a statin in the treatment of estrogen receptor positive breast cancer. Patients will take oral rosuvastatin daily. The maximum number of patients evaluable for a DLT is 12. Dosing will be as follows: Cohort 1 - rosuvastatin 20mg, Cohort 2 - rosuvastatin 40mg. The patients will have a total of 4 blood draws and 4 breast biopsies. The breast biopsies will be collected to evaluate cholesterol metabolites and tumor microenvironment characteristics including gene expression profiling and metabolomics. Sampling will occur at study entry, week 4, week 8, and at the time of surgery in early stage patients or at week 16 for metastatic patients. Patients will begin endocrine therapy following the acquisition of week 4 samples (blood and tissue biopsy).

ELIGIBILITY:
Inclusion Criteria:

* Women with ER+/PR+ HER2-negative breast cancer initiating neoadjuvant endocrine therapy with curative intent OR initiating endocrine therapy for the treatment of metastatic breast cancer with a biopsy accessible primary breast tumor
* The patients may start any FDA approved endocrine therapy (with which they have not been previously treated) at week 4 of the trial except for tamoxifen
* Palbociclib can be started at week 4, if indicated
* Patients with metastatic disease currently on endocrine therapy must be willing to stop endocrine therapy for 2 weeks prior to starting the study and to switch to a new endocrine therapy on the study (at week 4)
* Intact breast tumor present and size measuring at least 1cm at enrollment
* Post-menopausal at enrollment (age ≥ 60, age ≤ 60 and amenorrhea for ≥12 months in the absence of chemotherapy, tamoxifen, ovarian suppression and FSH/estradiol in the post-menopausal range)
* ECOG ≤ 2
* Can be on other endocrine therapy if willing to change a different endocrine therapy agent for the trial
* Must have at least one FDA approved endocrine therapy option with which the patient has not received prior treatment
* Life expectancy > 12 weeks
* Laboratory criteria: normal renal function: creatinine < 1.5 x upper limit of normal (ULN)), liver function: bilirubin < 2 x ULN, transaminases < 2 x ULN and blood counts: WBC ≥ 2.0, Neutrophils ≥1250, platelets ≥50,000, Hemoglobin ≥ 8.
* Age > 18 years
* Patients must have the ability to give informed consent.
* Patients must have a signed informed consent form prior to enrollment on study. -

Exclusion Criteria:

* Statin use in the last 6 months
* Patient has been treated with all FDA approved endocrine therapies or has been treated with all FDA approved endocrine therapies except for tamoxifen (tamoxifen is excluded from the trial)
* Active liver disease with elevated transaminases > 2x ULN
* Known hypersensitivity to rosuvastatin
* Any history of any other cancer (except non-melanoma skin cancer or carcinoma in-situ of the cervix) unless the patient has been in remission and off all other cancer therapy for at least 3 years.
* Patients should have no significant psychiatric illness or medical illness that would preclude the ability to comply with the protocol.
* Patients currently taking medications with known rosuvastatin interactions including cyclosporine, gemfibrozil, lopinavir/ritonavir, atazanavir/ritonavir, coumarin anticoagulants, colchicine, fenofibrates, and niacin.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2017-05-10 (Actual); Study Completion 2017-05-10 (Actual)

PRIMARY OUTCOMES:
Safety by adverse event | Neoadjuvant - 16 weeks prior to surgery
Maximum tolerated dose | Neoadjuvant - 16 weeks prior to surgery

SECONDARY OUTCOMES:
Change in Ki-67 with rosuvastatin alone followed by rosuvastatin in combination with endocrine therapy | 12 months after final tumor sample collection
progression free survival | 5 years after last subject completion

CONTACTS AND LOCATIONS:
Overall Officials: Kimberly Blackwell, M.D., Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States